CLINICAL TRIAL: NCT05830890
Title: A Clinical Trial of Sentinel Lymph Node Biopsy in Rectal Cancer
Brief Title: Sentinel Lymph Node Biopsy in Rectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Cancer Center, China (Other)
Responsible Party: Principal Investigator, Haitao Zhou, Clinical Professor, National Cancer Center, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SLNB
Record Dates: First submitted 2023-03-15; First posted 2023-04-26 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Rectal Cancer Stage III; Rectal Cancer Stage IV
Keywords: Laparoscope; Rectal cancer; Indocyanine green; Sentinel lymph node; lymph node dissection
MeSH Terms: conditions — Rectal Neoplasms | interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sentinel Lymph Node Biopsy (Experimental): The fluorescence laparoscope was used to visualize and locate the sentinel lymph node, which was then removed.
  Interventions: Procedure: Sentinel lymph node biopsy; Drug: Indocyanine green solution; Device: fluorescence laparoscope; Diagnostic Test: pathological examination; Diagnostic Test: rapid frozen pathological examination; Procedure: total mesorectal excision

INTERVENTIONS:
Procedure: Sentinel lymph node biopsy — After the total mesorectal excision, the indocyanine green was injected around the tumor via the anus. The fluorescence laparoscope was used to visualize and locate the sentinel lymph node, which was then removed and sent for rapid frozen pathological examination. Subsequently, a lateral lymph node dissection was performed.
  Other Names: Lateral lymph nodes dissection
Drug: Indocyanine green solution — Indocyanine green was injected around the tumor via the anus to visualize the sentinel lymph nodes under the fluorescence laparoscope.
  Other Names: Indocyanine green fluorescence imaging
Device: fluorescence laparoscope — The fluorescence laparoscope was used to visualize and locate the sentinel lymph node.
Diagnostic Test: pathological examination — The surgical specimens and sentinel lymph nodes were routinely examined for pathology.
Diagnostic Test: rapid frozen pathological examination — The lateral green fluorescence imaging sentinel lymph nodes found during surgery was sent to make cryosections. And then a pathologist makes a rapid diagnosis under a microscope。
Procedure: total mesorectal excision — 1. Sharply dissect the vascular interface between the pelvic fascia parietal layer and the visceral layer around the mesentery under direct vision to ensure that the rectal mesentery of the resected specimen is intact and tearless.
  2. For medium and low rectal cancer: the distal intestinal tube of the tumor should be resected ≥ 2 cm.
  3. TME or mesenteric distal resection margin ≥ 5 cm away from the tumor.
  Other Names: TME

SUMMARY:
Rectal cancer is one of the most common malignant tumors, with 9% to 23% of patients experiencing pelvic sidewall lymph node metastasis. According to the current Chinese guidelines for diagnosing and treating colorectal cancer, pelvic sidewall lymph node dissection is recommended for patients who have experienced or are suspected of having lateral lymph node metastasis. Lateral lymph node dissection can result in longer operation times, increased bleeding, and complications such as urinary and sexual dysfunction after surgery. Currently, the presence of metastasis is primarily determined by the size and enhancement characteristics of lateral lymph nodes observed through imaging studies. However, the pathological lymph node metastasis rate of specimens collected after lateral lymph node dissection based on current imaging criteria is only 20.5%. Therefore, a pressing clinical challenge is accurately determining the presence of lateral lymph node metastasis and avoiding unnecessary lateral lymph node dissection in patients who have not experienced lateral lymph node metastasis.

Sentinel lymph node biopsy has been widely used in clinical practice. It has replaced traditional lymph node dissection in some breast cancer and melanoma patients, reducing surgical risks and complications and improving patients' quality of life. This study aims to use indocyanine green as a tracer for fluorescence-guided laparoscopic navigation to locate the lateral sentinel lymph nodes of rectal cancer in the pelvic cavity. By studying the accuracy, specificity, and false-negative rate of predicting lateral lymph node status using the sentinel lymph node, we can further clarify the clinical significance of the lateral sentinel lymph node.

DETAILED DESCRIPTION:
This study is a prospective single-arm clinical study. 87 patients with middle and low rectal cancer are planned to be included in the study. After general anesthesia during the operation, indocyanine green is injected around the tumor through the anus. After the sentinel lymph nodes are developed and located by fluorescent laparoscopy, they are removed and sent to rapid frozen pathological examination, and then the lateral lymph nodes are cleaned. Through pathological examination and statistical analysis of the fluorescent stained lateral sentinel lymph nodes and all the cleaned lateral lymph nodes, To evaluate the clinical significance of lateral sentinel lymph nodes located by this technique in predicting the status of lateral lymph nodes.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 75 years old.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0-1.
* Newly diagnosed patients with confirmed rectal cancer by histopathology.
* Preoperative clinical staging by imaging examination is T3-4.
* Preoperative colonoscopy shows the distance from the tumor's lower edge to the anus is less than 10cm.
* No previous chemotherapy or radiotherapy.
* Preoperative imaging examination (pelvic enhanced MRI) shows lateral lymph nodes with a maximum short diameter of ≥5mm and <10mm.
* Women of childbearing age must take effective contraceptive measures.
* Able to understand the study and sign the informed consent form.

Exclusion Criteria:

* Complete intestinal obstruction.
* Active hepatitis and peripheral neuropathy (such as peripheral neuritis, pseudomeningitis, motor neuritis, sensory disturbances, etc.).
* Pregnant or lactating women; women of childbearing potential who have not taken sufficient contraceptive measures.
* History of other tumors or previous chemotherapy or radiotherapy.
* Alcoholism or drug addiction.
* Significant organ dysfunction or other significant diseases, including clinically relevant coronary artery disease, cardiovascular disease, or myocardial infarction within 12 months before enrollment; severe neurological or psychiatric history; severe infection; active disseminated intravascular coagulation.
* Hypoproteinemia.
* Preprandial blood glucose control exceeds 11.2mmol/L in the week before surgery.
* BMI>28 kg/m^2.
* Poor compliance, and failure to comply with the study protocol.
* Subject withdrawal from the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
False negative rate | up to 14 days
  The false negative rate of predicting lateral lymph node metastasis status using rapid frozen pathology results of lateral sentinel lymph nodes in mid-to-low rectal cancer.
  Namely, the false negative rate= total false negative cases/(total false negative cases+total true positive cases).
Accuracy | up to 14 days
  The accuracy of predicting lateral lymph node metastasis status using rapid frozen pathology results of lateral sentinel lymph nodes in mid-to-low rectal cancer.
  Namely, the accuracy = (total true negative cases+total true positive cases)/total number of cases.

SECONDARY OUTCOMES:
Detection rate | up to 14 days
  The detection rate of lateral sentinel lymph nodes in middle and low rectal cancer.
  Namely, the detection rate = (total true positive cases+total false positive cases)/total number of cases.
Specificity | up to 14 days
  The specificity of predicting lateral lymph node metastasis status using rapid frozen pathology results of lateral sentinel lymph nodes in mid-to-low rectal cancer.
  Namely, the specificity = total true negative cases/(total true negative cases+total false positive cases).
Sensitivity | up to 14 days
  The Sensitivity of predicting lateral lymph node metastasis status using rapid frozen pathology results of lateral sentinel lymph nodes in mid-to-low rectal cancer.
  Namely, the sensitivity= total true positive cases/(total true positive cases+total false negative cases)。

CONTACTS AND LOCATIONS:
Overall Officials: Haitao Zhou, M.D., Study Chair — National Cancer Center, China
Locations (1):
- National Cancer Center, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Participants' data are only allowed to be used for the analysis of this study and are not authorized to be shared with other researchers.